CLINICAL TRIAL: NCT00178347
Title: Radiation Dosimetry in Teeth
Status: Terminated | Type: Observational
Sponsor: University of Rochester (Other)
Responsible Party: Paul Okunieff, University of Rochester, Medical Center
Other Study IDs: URCC 11070
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2009-05-19 (Estimated); Status verified 2009-05

CONDITIONS: Radiation Tolerance

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Radiation: Exposure to irradiation — Treatment for Cancer using Radiation -dose will be the standard of Care for the type of Cancer being treated

SUMMARY:
Irradiation of any tissue creates changes in that tissue. Ionizing radiation imparts charges to the tissue as it interacts with tissue components, changing the tissue structure. The specific type of modification also depends to some extent upon the type of tissue irradiated. It has been shown that it is possible to read the tooth enamel irradiation record using techniques such as electron paramagnetic resonance (EPR), or electron spin resonance (ESR).

It is proposed to examine radiation responses in approximately one hundred (100) human teeth. This would include teeth free of, as well as those containing, amalgam (silver) restorations. For the first group, teeth that have already been collected (pre-existing pathological specimens) would be used. These teeth were surgical/pathological discards collected without identifiers by the dental providers.

ELIGIBILITY:
Inclusion Criteria:

* Discarded pathologic specimens (teeth)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: discarded pathological specimen(teeth)
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2004-12

CONTACTS AND LOCATIONS:
Overall Officials: Paul Okunieff, MD, Study Chair — University of Rochester, Dept. of Radiation Oncology
Locations (1):
- University of Rochester, Dept. Radiation Oncology, Rochester, New York, United States